CLINICAL TRIAL: NCT06250140
Title: A Multicenter Retrospective Study on the Recurrence Rate of Minimally Invasive Endoscopic Treatment of Internal Hemorrhoids
Brief Title: Recurrence Rate of Minimally Invasive Endoscopic Treatment of Internal Hemorrhoids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Collaborators: 964 hospital of joint Logistics Support Force (Unknown); The Chinese people's liberation army army medical center (Unknown)
Responsible Party: Principal Investigator, Ying Zhu, Professor, Shenzhen Hospital of Southern Medical University
Other Study IDs: ShenzhenH
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Internal Hemorrhoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Internal hemorrhoid ligation group: Endoscopic internal hemorrhoid ligation
  Interventions: Device: Tie up device
- Hemorrhoids injection group: Endoscopic hemorrhoid injection was performed
  Interventions: Device: Tie up device
- Internal hemorrhoids combined treatment group: Lines of endoscopic hemorrhoids and internal ligation under endoscope to injection
  Interventions: Device: Tie up device

INTERVENTIONS:
Device: Tie up device — The recurrence rate of internal hemorrhoids in different treatment methods

SUMMARY:
2.1 Main objective: To observe the short-term and long-term recurrence rates of various endoscopic minimally invasive treatment methods for internal hemorrhoids and different time points of endoscopic minimally invasive treatment for internal hemorrhoids in patients with grade I-III internal hemorrhoids

2.2 Secondary objective: To observe the safety and efficacy of endoscopic minimally invasive treatment of internal hemorrhoids

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, both sexes

  2, grade I-III internal hemorrhoids with symptoms related to internal hemorrhoids

  3. The purpose and adverse consequences of endoscopic minimally invasive treatment of internal hemorrhoids have been fully understood before surgery, and the informed consent for endoscopic minimally invasive treatment of internal hemorrhoids has been signed

Exclusion Criteria:

* 1. Patients with contraindications to endoscopic minimally invasive treatment (1) grade IV internal hemorrhoids, mixed hemorrhoids and external hemorrhoids; (2) I-III

Degree of internal hemorrhoids with incarceration, thrombosis, erosion, infection, etc. (3) patients with severe systemic diseases could not tolerate endoscopic treatment; (4) accompanied by crissum infectious disease, anal fistula, and inflammatory bowel disease activity, etc.; (5) in menstrual period, pregnancy and puerperium, (6) patients with sclerotherapy allergy; (7) function of blood coagulation disorder or are using anticoagulant drugs.

2. Patients with a history of allergy to narcotic drugs

3. Patients who were deemed by the investigator to be ineligible for participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with internal hemorrhoids who had undergone endoscopic treatment for internal hemorrhoids could be enrolled in the study after informed consent was obtained
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of minimally invasive endoscopic treatment | One year
  If patients with internal hemorrhoids recurred with preoperative clinical symptoms (bleeding, prolapse, pain, etc.), which could not be relieved by conservative treatment, and needed endoscopic sclerotherapy, ligation, ligation sclerotherapy or surgery again, the recurrence rate = the number of recurrent cases/the number of patients X100%

SECONDARY OUTCOMES:
The overall efficacy of various treatment methods | One year
  (1) Cure: the symptoms of hematochezia and prolapse disappeared completely. (2) Remarkable effect: the symptoms of hematochezia and prolapse were significantly improved, or the symptoms were alleviated but the frequency and degree of attack were reduced compared with those before operation; (3) Ineffective: the symptoms of hematochezia and prolapse were not relieved or even aggravated. Total effective rate = (cure + marked effective)/total ratio X100%
Recurrence rates of various treatment modalities in different grades | One year
The efficacy of sequential treatment after recurrence was evaluated | One year
  Patients with internal hemorrhoids who had preoperative clinical symptoms (bleeding, prolapse, pain, etc.) at more than 3 months after operation, and failed to be relieved by conservative treatment, needed endoscopic sclerotherapy, ligation, ligation sclerotherapy or surgery again were regarded as recurrence. Total effective rate = (cure + marked effective)/total ratio X100%

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT06250140/ICF_000.pdf